CLINICAL TRIAL: NCT04340986
Title: Cohort Study of Patients With Primary Hepatocellular Carcinoma or Cholangiocarcinoma
Brief Title: Cohort of Patients With Hepatocellular Carcinoma or Cholangiocarcinoma
Acronym: CHC/CC
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP190473; IDRCB 2019-A01679-48 (Other: ANSM)
Record Dates: First submitted 2020-04-07; First posted 2020-04-10 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Cholangiocarcinoma; Hepatocellular Carcinoma
Keywords: hepatocellular carcinoma; cholangiocarcinoma; cohort
MeSH Terms: conditions — Cholangiocarcinoma; Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with Hepatocellular carcinoma
- patients with Cholangiocarcinoma

SUMMARY:
The main objective is to describe the evolution of patients treated for a primary malignant hepatobiliary tumor (hepatocellular carcinoma or cholangiocarcinoma) over the long course.

DETAILED DESCRIPTION:
The collection of data from patients with CHC and cholangiocarcinomas who are cancers with poor prognosis is a major challenge to improve patients'care (diagnosis, prognosis); facilitate the search for new therapeutic targets and the follow-up of clinical studies; and develop personalized treatments.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria :

* Age ≥ 18 years olds
* Medical care in Nephrology department since 2015

Cholangiocarcinoma:

- Histologically and cytologically documented cholangiocarcinoma, regardless of the stage of the disease

Hepatocellular carcinoma:

* Hepatocellular carcinoma at any stage of the disease, presenting the diagnostic criteria according to the diagnostic criteria of Barcelona : Tumor of more than 1 cm, developed on cirrhosis liver with arterial phase hyperenhancement and washout in the portal venous or delayed phases on CT and MRI
* Hepatocellular histologically documented

Exclusion Criteria:

- Lack of patient non-opposition

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients with hepatocellular carcinoma or cholangiocarcinoma treated in Saint-Antoine hospital
Sampling Method: Probability Sample
Enrollment: 1250 (Estimated)
Dates: Start 2020-09-02 (Actual); Primary Completion 2030-09 (Estimated); Study Completion 2030-09 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 5 years
  Hepatocellular carcinoma and Cholangiocarcinoma : Overall survival is defined as the survival 5 years after the inclusion.

SECONDARY OUTCOMES:
Overall survival | 5 years
  Hepatocellular carcinoma :Overall survival is defined as the survival after 5 years of inclusion.
Disease free survival | 2 and 5 years
  Cholangiocarcinoma : 2 and 5 years after surgical resection
Progression time under chemotherapy | Time of progression under chemotherapy up to 5 years
  Cholangiocarcinoma : Time of progression under chemotherapy is defined by the delay between the start of chemotherapy and tumor progression (appearance of a new lesion or increase in size of more than 30%)

CONTACTS AND LOCATIONS:
Overall Officials: Marie LEQUOY, MD, Principal Investigator — AssistancePublique-Hôpitaux de Paris
Locations (1):
- Serviec hépatologie-Hôpital Saint Antoine, Paris, France

IPD SHARING:
Plan to Share IPD: No